CLINICAL TRIAL: NCT02760628
Title: A Clinic and Tech-Based Diet and Fitness Intervention for Volunteer Firefighters
Brief Title: The First Twenty (TF20) for Volunteer Firefighters in a Clinic Based Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R34HL125790-01 (NIH)
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The First Twenty (TF20) (Experimental): Participants in TF20 will be provided an online wellness program focused on fitness and nutrition tailored to firefighters. TF20 is interactive and involves health coaching.
  Interventions: Behavioral: The First Twenty (TF20)
- Life Simple Seven (LS7) (Placebo Comparator): Participants assigned to the LS7 arm will be directed to a website that contains information about health and wellness from the American Heart Association that was developed for the general population. No health coaching is present and the site is not tailored for the fire service.
  Interventions: Behavioral: Life Simple 7 (LS7)

INTERVENTIONS:
Behavioral: The First Twenty (TF20) — TF20 is an online wellness program for firefighters focused on improving cardiovascular risk factors through behavioral changes.
  Arms: The First Twenty (TF20)
Behavioral: Life Simple 7 (LS7) — LS7 is a wellness program designed and implemented by the American Heart Association focused on improving cardiovascular health.
  Arms: Life Simple Seven (LS7)

SUMMARY:
The First Twenty® (TF20) was recently developed as a not-for-profit, web-mobile program for firefighters (FFs) specifically focused on improving fitness and nutrition knowledge and practices. The program was designed by FFs with backgrounds in tactical fitness, marketing and program development professionals, and nutrition and exercise scientists. Preliminary data suggests the program is well-received by FFs and results in significant improvement in body composition and physical fitness. One innovative approach for the eventual dissemination of TF20 to VFFs is through their fitness-for duty medical exams. The synergy created by linking the TF20 intervention components, feedback to the VFFs from their medical exam, and health messages from their physician is predicted to maximize the impact of this much-needed intervention. The goal of the proposed project is to tailor TF20 for use in a clinic based setting (CB-TF20) for VFFs and to pilot test it in comparison to the American Heart Association's Life's Simple 7 (LS7), a web-based diet and physical activity knowledge/behavior and lifestyle program. The specific aims are to: 1) Conduct formative research with key stakeholders in the VFF community (e.g., physicians, department leadership, VFFs) to determine best practices for implementing a clinic-based, web-mobile health and wellness program with VFFs and medical providers; 2) Develop a clinic-based version of TF20 (CB-TF20) and beta-test it with VFFs; and, 3) Conduct a 6 month, 2-arm, pilot cluster (i.e., department) randomized clinical trial (PCRCT) to determine the comparative effectiveness of the revised CB-TF20 to LS7 on body composition, Framingham Risk Scores, and diet/physical activity knowledge and behaviors among VFF with BMI >25.0kg/m2; and conduct an evaluation of the CB-TF20 materials and technology. This innovative R34 study is a critical step in providing a much needed intervention for VFFs and those providing their annual examinations.

DETAILED DESCRIPTION:
The US fire service serves as the front line of defense against any domestic emergency and volunteer firefighters comprise the majority of firefighters, often with negative consequences for the health of personnel. While rates of overweight and obesity remain high among firefighters and cardiovascular disease remains the leading cause of line of duty deaths, few resources tailored to the unique culture and needs of firefighters are available to help occupational medicine physicians who provide their fitness for duty examinations. By engaging firefighters and occupational medicine clinicians in tailoring an internet/mobile intervention and pilot testing the program with a sample of volunteer firefighters, the investigators will be poised to implement a full-scale clinical trial with the developed program.

ELIGIBILITY:
Inclusion Criteria:

* Willing to complete all assessments
* Internet accessibility via computer, tablet or smartphone and ability to use devices appropriately
* Medically cleared to participate in the program through clinicians
* ≥18 years

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Body Fat | 6 months
  Body fat as measured by foot-to-foot bio-electrical impedance

SECONDARY OUTCOMES:
Framingham Risk Score | 6 months
Body Mass Index (BMI) | 6 months
  BMI as calculated by weight in kilograms/height in meters squared
Waist circumference | 6 months
  Waist circumference as measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Sara Jahnke, PhD, Principal Investigator — National Development & Research Institutes
Locations (2):
- United States (2):
  - NDRI Institute of Bioebehavioral Health Research, Leawood, Kansas
  - National Development and Research Institutes, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided